CLINICAL TRIAL: NCT01890135
Title: A Phase II Clinical Trail to Assess the Safety and Effects of ZD4054 (Zibotentan) on Exercise Induced Calf Muscle Perfusion in Patients With Intermittent Claudication (Rutherford II or III).
Brief Title: Zibotentan, an Endothelin Receptor Antagonist, Patients With Intermittent Claudication
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Brian Annex, MD, Professor of Medicine, Chief Division of Cardiovascular Medicine, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 17030
Record Dates: First submitted 2013-06-18; First posted 2013-07-01 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-08

CONDITIONS: Peripheral Arterial Disease; Intermittent Claudication
Keywords: randomized; double blind; blood flow; muscle perfusion; safety
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication | interventions — ZD4054

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- endothelin receptor antogonist (Active Comparator): 10 mg of zibotentan
  Interventions: Drug: Zibotentan (ZD4054); Drug: placebo
- placebo (Placebo Comparator): matched placebo
  Interventions: Drug: Zibotentan (ZD4054); Drug: placebo

INTERVENTIONS:
Drug: Zibotentan (ZD4054) — 10 mg
Drug: placebo — randomized double blind
  Other Names: matched placebo

SUMMARY:
Peripheral artery disease (PAD) is a major complication of atherosclerosis when blockages in the arteries to leg reduce blood flow and one of the resulting problems is termed intermittent claudication (IC). IC is leg pain with walking that is relieved with rest and IC is the most frequent clinical manifestation of PAD and it effects millions of Americans. The number of patients with, and the health care costs of, PAD will increase as the prevalence of PAD is associated with advancing age, diabetes, and smoking. Zibotentan (ZD4054) is an endothelin receptor A (ETA) blocker that undergone extensive human testing and has been shown to be safe in several patient population. There is ample evidence to suggest that an ETA blocker could improve blood flow to the legs in patients with PAD. In a study that will be funded by the National Institute of Health, the investigators will test the ability of this medication to allow better blood flow to the legs of patients with PAD. In patients with IC, the investigators will test the ability of ZD4054 to improve leg blood flow using a non-invasive imaging technique. In parallel the study will test for the ability of patients with leg pain to walk further and feel better.

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) is a major complication of atherosclerosis that affects >8 million people in the United States alone. Intermittent claudication (IC), defined as leg pain with walking that is relieved with rest, is the most frequent clinical manifestation of PAD.

In a proposal that was just funded by the National Institute of Health (NIH) National Center for Advancing TRanslational Sciences (NCATS) the investigators pose to test the "reuse" of zibotentan (ZD4054, an Asta-Zeneca compound), an orally active, endothelin receptor A (ETA) antagonist in patients with IC. The study will seek to confirm the safety and tolerability of 10mg of ZD4054 in patients with intermittent claudication (Rutherford II or III) and, in parallel, establish the capacity of ZD4054 to change calf muscle perfusion, as assessed by contrast-enhanced magnetic resonance imaging, functional treadmill performance, and quality of life indicators.

The study will be a 1:1 randomized, double-blind, placebo-controlled trial of 44 subjects with intermittent claudication with randomization stratified based on the entry calf muscle perfusion. The investigators will use magnetic resonance imaging to quantify changes in blood flow to the ischemic limb from baseline to week 12 between those randomized to drug vs. placebo. Based on the prior experience and the known tolerability of ZD4054, the experience of the investigative team with a mechanistically appropriate end-point measure that is part of other NIH funded projects, the investigators will proceed directly to this Phase II trial. The primary endpoint of the study will be the change in absolute perfusion in the index calf muscle from baseline to follow-up, after 12 weeks on the 10 mg dose or placebo. Additional outcome measures will be: a) ability of patients with PAD to tolerate 10 mg dose of ZD4054 vs. placebo; b) freedom from unexpected serious adverse events; c) change in peak walking time from baseline to 12 weeks between 10 mg of ZD4054 and placebo groups; d) change in ankle-brachial blood pressure index (ABI) from baseline to 12 weeks between 10 mg of ZD4054 and placebo groups, and; d) change in quality of life measure between 10 mg of ZD4054 and placebo groups.

ELIGIBILITY:
Inclusion Criteria:

* Age >40 years. Patients less than 40 years of age could well have a form or "thromboangitis obliterans" often called Berger's Disease and the investigators wish to enroll only subjects with atherosclerotic vascular disease.
* Currently taking all standard medications that are part of the "good medical care" for patients with PAD including an anti-platlet agent, an angiotensin-converting enzyme inhibitors or receptor blockers, beta-blockers if indicated for ischemic heart disease, and cholesterol lowering therapy; unless documented contra-indications to these therapies exist. Those patients not on these therapies will be referred back with the suggestion that they be added and they can be re-approached for enrollment at a later date.
* Exercise induced thigh, calf, buttock pain and absence of Rutherford Class IV, V, or VI.3
* A resting ABI of <0.9 but >0.4 and the presence of both superficial femoral artery stenosis (70% or greater) disease and below the knee disease with a significant stenosis in at least one of the run-off vessels.
* Absence of critical inflow (iliac or common femoral) disease. The profunda femoral artery is the major source of collateral blood vessels. The investigators initial approach will be to try and enroll as homogenous of a patient population as possible to allow us to focus on the primary endpoint of the study (the change in muscle perfusion to the ischemic limb over time).
* Ability to undergo magnetic resonance imaging and provide informed written consent.

Exclusion Criteria:

* Serious known concomitant disease with life expectancy of less than one year
* Prior amputation or history of critical limb ischemia
* Creatinine clearance (CrCl) >45 to permit safe administration of the gadolinium contrast agent.
* Recent myocardial infarction, unstable angina, stroke or transient ischemic attack within 3 months.
* American Heart Association Class III or IV congestive heart failure or known left ventricular ejection fraction less than 40%.
* Known history of anemia

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in exercise-induced calf muscle perfusion by magnetic resonance imaging | Baseline and 12 weeks

SECONDARY OUTCOMES:
Change in peak walking time | Baseline and 12 weeks
  Peak walking time (PWT) will be measured using the Gardner treadmill protocol which is designed for patients with peripheral arterial disease.
Change in quality of life measures | Baseline and 12 weeks
  Quality of life measures specific to peripheral arterial disease will be assessed by questionnaire.
Safety | Baseline and Day 30
  Confirmation of lack of change in edema or heart failure by history and physical examination

OTHER OUTCOMES:
Change in ankle-brachial blood pressure index (ABI | Baseline and 12 weeks
Change in hematocrit | baseline and day 30

CONTACTS AND LOCATIONS:
Overall Officials: Brian H Annex, MD, Principal Investigator — University of Virginia
Locations (1):
- University Of Virginia Health System, Charlottesville, Virginia, United States